CLINICAL TRIAL: NCT00343928
Title: Amino Acids, Serotonin, and Body Weight Regulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2004P000107; R21MH071689 (NIH); 2004P-000107 DATR A2-AID
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Branched-chain amino acids

INTERVENTIONS:
Other: Branched-chain amino acids — Participants will spend approximately 2 weeks in each phase over a 9-week period, during which they will receive an amino acid mixture and the placebo control condition.

SUMMARY:
This study will assess the behavioral effects of an amino acid mixture thought to influence serotonin function in individuals who have recovered from anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa is a serious psychiatric disorder resulting in psychosocial distress for patients and their families, potentially severe medical consequences, and substantial long-term mortality. A major emphasis in current therapeutic research in anorexia nervosa is exploration of new interventions to stabilize recovery and prevent relapse. Although the etiology of anorexia nervosa is unknown, altered regulation of the neurotransmitter serotonin in the central nervous system is thought to contribute to preoccupation with body shape and weight, dysregulated eating patterns, persistent anxiety, and frequent mood fluctuations. The goal of this exploratory project is to assess the behavioral effects of an amino acid mixture thought to influence serotonin function in individuals who have recovered from anorexia nervosa. It is hypothesized that this brief intervention will help diminish residual eating disorder symptoms.

All participants in this crossover study will attend eight sessions over a 9-week period. Participants will spend approximately 2 weeks in each phase, during which they will receive an amino acid mixture and the control condition.

ELIGIBILITY:
Inclusion Criteria:

* History of anorexia nervosa
* In normal weight range with resumed menses
* No recent bulimic episodes
* Persistent symptoms of anxiety

Exclusion Criteria:

* Currently treated with psychotropic medication
* Diagnosed with major depression
* Current or recent substance dependence
* Serious medical illness
* Pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Anxiety and preoccupation with body image | Measured at Week 9

SECONDARY OUTCOMES:
Eating patterns | Measured at Week 9

CONTACTS AND LOCATIONS:
Overall Officials: David C. Jimerson, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States